CLINICAL TRIAL: NCT01392118
Title: Recurrent ESBL-producing Enterobacteriaceae Bacteremia: Risk Factor, Molecular Character and Susceptibility Change
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Chen-Hsiang Lee / Chief; Division of Infectious Diseases, Chang Gung Medical Foundation, Kaohsiung Branch
Other Study IDs: MISP38634
Record Dates: First submitted 2011-07-10; First posted 2011-07-12 (Estimated); Last update posted 2011-07-12 (Estimated); Status verified 2011-01

CONDITIONS: Bacteremia
MeSH Terms: conditions — Bacteremia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — ESBL strains of E. coli or K. pneumoniae from blood cultures under normal practice
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to investigate the risk factor, molecular character and susceptibility change for recurrent ESBL-producing Enterobacteriaceae bacteremia

DETAILED DESCRIPTION:
1. To characterize the genotypes of the pathogens isolated from recurrent ESBL-EK bacteremia versus non-recurrent ESBL-EK bacteremia to differentiate relapse from reinfection

   * recurrent versus non-recurrent
   * relapse versus reinfection
2. To correlate the patient characteristics, clinical manifestations, severity of illness (the modified Pitt bacteremia score), diagnosis of deep-site infection, co-morbid conditions (including diabetes mellitus, hepatic and renal dysfunction), length of stay in ICU/hospitalization, the presence of invasive procedures, source of pathogen (community acquired or nosocomial infection), antimicrobial regimen (i.e carbapenems versus non-carbapenems(flomoxef or quinolones), microbiological characteristics (E coli and Kleb. pneumoniae) and outcome endpoints (clinical outcome and mortality) with ESBL recurrence and genotypes

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age>=18 years) with at least one episode of ESBL-EK bloodstream infection from August 2004 to July 2010

Exclusion Criteria:

* Patients who died within 48h after first episode of ESBL-EK bloodstream infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In a tertiary care hospital, every adult patient with at least one episode of ESBL-EK bloodstream infection from August 2004 to July 2010 will be recruited into this study. Patients who died within 48h after first episode of ESBL-EK bloodstream infection will be excluded.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2011-07; Study Completion 2012-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Chen-Hsiang Lee, M.D., Principal Investigator — Chang Gung Medical Foundation, Kaohsiung Branch
Locations (1):
- Chang Gung Medical Foundation, Kaohsiung Branch, Kaohsiung City, Taiwan